CLINICAL TRIAL: NCT02041741
Title: Happiness in Flanders: A Randomized, Wait-List Controlled Study
Brief Title: Improving Happiness in Flanders
Acronym: HAP-FLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAP-FLA
Record Dates: First submitted 2014-01-13; First posted 2014-01-22 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2014-01

CONDITIONS: Happiness in the General Population
Keywords: happiness; well-being; distress; positive psychology

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Weekly tips (Active Comparator): Daily small and concrete happiness tips
  Interventions: Behavioral: Weekly tips
- Daily Tips (Active Comparator): Weekly more in-depth happiness tips involving an active (doing and experiencing) task
  Interventions: Behavioral: Daily Tips
- Wait-List Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Weekly tips — Participants in this condition receive weekly a more in-depth tip to increase feelings of happiness involving a (doing and experiencing) task
  Arms: Weekly tips
Behavioral: Daily Tips — Participants in this condition receive daily a set of small tips aimed at increasing happiness
  Arms: Daily Tips

SUMMARY:
This study aims to assess the effects of two different types of interventions aimed at increasing happiness in the Flemish general population as compared to individuals that receive no intervention.

DETAILED DESCRIPTION:
This randomized trial has two aims:

1. First, it investigates the efficacy of two different happiness interventions in increasing feelings of happiness in the Flemish general population using a wait-list controlled design.
2. Second, this study aims to identify predictors of response in both interventions ("what works for whom?")

Methods

Design and procedure

* Participants will be contacted through social media and directed to a website that is specifically designed for this study.
* All participants who register for the study first will electronically sign an informed consent and will be asked to complete a brief battery of questionnaires online (base line measures) before randomization.
* Participants then are assigned randomly using a block-randomized design to one of the three conditions using a computerized algorithm:

  1. a condition in which daily small and concrete happiness tips are sent to participants during one month via email (n=400)
  2. a condition in which weekly more in-depth happiness tips with a (doing and experiencing) task are given during one month via email (n=400)
  3. a wait-list condition (1 month); these participants will be subsequently (after the end of the 4-week intervention) randomized to condition (a) or (b) (n=400) using a block-randomized design.
* All participants will be assessed weekly during the intervention (see below) and followed-up 6 months after the end of the study.

Measures

Participants will complete a detailed demographic questionnaire.

Primary outcome measures:

* Subjective Happiness Scale (SHS; Lyubomirsky & Lepper, 1999)
* Steen Happiness Inventory (SHI; Seligman, Steen, Park, & Peterson, 2005)

Secondary outcome measures

* Positive and Negative Affect Scales (PANAS; Watson, Clark, & Tellegen, 1988)
* Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001)
* Warwick Edinburgh Mental Well-Being Scale (WEMWBS; Tennant et al., 2007)
* Brief Symptom Inventory (Korte KlachtenLijst; KKL; Lange, & Appelo, 2007)

Predictors of outcome

* Meaning in Life Questionnaire (MLQ; Steger, Frazier, Oishi, & Kaler, 2006)
* Depressive Experiences Questionnaire (DEQ; Blatt, D'Afflitti, & Quinlan, 1976)
* Experiences in Close Relationships-Revised (ECR-R, Fraley, Waller, & Brennan, 2000)
* Kentucky Inventory of Mindfulness (KIMS; Baer, Smith, & Allen, 2004)
* Toronto Alexithymia Scale (TAS; Bagby, Parker, & Taylor, 1994)

Data analyses

Repeated measures Anova and multilevel modeling will be used to assess differences between the three conditions in primary and secondary outcomes at the end of the intervention and at follow-up. Regression analyses and growth curve modeling will be used to examine the effects of the predictors on primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient fluency in Flemish
* at least 18 years of age

Exclusion Criteria:

* no fluency in Flemish
* living outside of Flanders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10863 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Subjective Happiness Scale | 4 weeks after start of intervention and 6 months after end of intervention
Steen Happiness Inventory | 4 weeks after start of intervention and 6 months after end of intervention

SECONDARY OUTCOMES:
Positive and Negative Affect Scale (PANAS) | 4 weeks after start of intervention and 6 months after end of intervention
Patient Health Questionnaire-9 (PHQ-9) | 4 weeks after start of intervention and 6 months after end of intervention
Warwick Edinburgh Mental Well-Being Scale | 4 weeks after start of intervention and 6 months after end of intervention
Brief Symptom Inventory (KKL, Korte KlachtenLijst) | 4 weeks after start of intervention and 6 months after end of intervention

OTHER OUTCOMES:
Meaning in Life Questionnaire | Start of intervention (predictor variable)
Depressive Experiences Questionnaire (DEQ) | Start of intervention (predictor variable)
Experiences in Close Relationships-Revised (ECR-R) | Start of intervention (predictor variable)
Kentucky Inventory of Mindfulness (KIMS) | Start of intervention (predictor variable)
Toronto Alexithymia Scale (TAS) | Start of intervention (predictor variable)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Luyten, PhD, Principal Investigator — KULeuven, Belgium; Mia Leijssen, PhD, Study Director — KULeuven, Belgium; Sara Casalin, PhD, Study Director — KULeuven, Belgium; Jessie Dezutter, PhD, Study Director — KULeuven, Belgium
Locations (1):
- Faculty of Psychology and Educational Sciences, Leuven, Belgium

REFERENCES:
- [Background] Seligman ME, Steen TA, Park N, Peterson C. Positive psychology progress: empirical validation of interventions. Am Psychol. 2005 Jul-Aug;60(5):410-21. doi: 10.1037/0003-066X.60.5.410. PMID 16045394
- [Background] Lyubomirsky, S., & Lepper, H. S. (1999). A measure of subjective happiness: Preliminary reliability and construct validation. Social Indicators Research, 46, 137-155.
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Blatt SJ, D'Afflitti JP, Quinlan DM. Experiences of depression in normal young adults. J Abnorm Psychol. 1976 Aug;85(4):383-9. doi: 10.1037//0021-843x.85.4.383. No abstract available. PMID 956505
- [Background] Fraley RC, Waller NG, Brennan KA. An item response theory analysis of self-report measures of adult attachment. J Pers Soc Psychol. 2000 Feb;78(2):350-65. doi: 10.1037//0022-3514.78.2.350. PMID 10707340
- [Background] Bagby RM, Parker JD, Taylor GJ. The twenty-item Toronto Alexithymia Scale--I. Item selection and cross-validation of the factor structure. J Psychosom Res. 1994 Jan;38(1):23-32. doi: 10.1016/0022-3999(94)90005-1. PMID 8126686
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Lange, A., & Appelo, M. (2007). Handleiding Korte Klachten Lijst (KKL) [Manual for the Brief Symptom Inventory]. Houten, The Netherlands: Bohn Stafleu Van Loghum.
- [Background] Steger, M. F., Frazier, P., Oishi, S., & Kaler, M. (2006). The Meaning in Life Questionnaire: Assessing the presence of and search for meaning in life. Journal of Counseling Psychology, 53(1), 80-93. doi: 10.1037/0022-0167.53.1.80
- [Background] Baer RA, Smith GT, Allen KB. Assessment of mindfulness by self-report: the Kentucky inventory of mindfulness skills. Assessment. 2004 Sep;11(3):191-206. doi: 10.1177/1073191104268029. PMID 15358875